CLINICAL TRIAL: NCT02695745
Title: Randomized, Double Blind, Positive- Controlled, Three-way Cross-over Human Experimental Biomarker Study of V116517 in Healthy Male Subjects
Brief Title: Experimental Biomarker Study for Pain Thresholds
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VND1004; 2011-002399-18 (EudraCT Number)
Record Dates: First submitted 2016-02-22; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Celecoxib; Capsaicin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- V116517 (Experimental): V116517 aqueous suspension; 300 mg
  Interventions: Drug: V116517 aqueous suspension; Drug: Placebo; Drug: Capsaicin
- Celecoxib (Active Comparator): Celecoxib capsules; 400 mg (2 capsules of 200 mg each)
  Interventions: Drug: Celecoxib capsules; Drug: Placebo; Drug: Capsaicin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo; Drug: Capsaicin

INTERVENTIONS:
Drug: V116517 aqueous suspension — 300 mg (approximately 100 mL) aqueous suspension taken orally x 1 dose
  Arms: V116517
Drug: Celecoxib capsules — 400 mg (2 capsules of 200 mg each) taken orally x 1 dose
  Other Names: Celebrex®; Celebra®
  Arms: Celecoxib
Drug: Placebo — Placebo for V116517 aqueous suspension taken orally x 1 dose and/or placebo for celecoxib, 2 capsules taken orally x 1 dose
Drug: Capsaicin — 1% administered topically

SUMMARY:
The purpose of this study is to characterize the heat pain tolerance threshold (HPTolTr) in primary hyperalgesic skin after topical capsaicin application, and to assess heat pain and mechanical thresholds (eg, pressure pain, stimulus-response) following skin sensitization by UVB (ultraviolet B) irradiation and topical capsaicin.

ELIGIBILITY:
Inclusion Criteria include:

1. Signed informed consent obtained.
2. Males aged 18 to 45, inclusive.
3. Body weight ranging from 50 to 100 kg and BMI ranging from 18 to 32 (kg/m2), inclusive.
4. Healthy and free of significant abnormal findings as determined by medical history, physical examination, clinical laboratory values, vital signs, and ECG.

Exclusion Criteria include:

1. Current or recent (within 5 years) history of drug or alcohol abuse.
2. History or any current conditions that might interfere with drug absorption, distribution, metabolism or excretion.
3. Any history of frequent nausea or emesis regardless of etiology.
4. Any history of allergic-type reactions to sulfonamides, or any experience of asthma, urticarial, or other allergic-type reactions after taking aspirin or other NSAIDS.
5. Subjects who do not develop erythema at the maximum dose of the UVB source (MED determination for UVB model) will be excluded from the study.

Other protocol-specific inclusion/exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Heat pain tolerance threshold (HPTolTr) in primary hyperalgesic skin after topical capsaicin application | 3.5 hours post-dose
  Mean temperature in degrees Celsius (°C) based on the difference (post-dose and pre-dose) of the differences between the capsaicin at the control arm and the treated arm

SECONDARY OUTCOMES:
Heat Pain Threshold (HPTr) | 3.5 hours post-dose
  Mean temperature in degrees Celsius (°C)
Heat Pain tolerance threshold (HPTolTr) | Pre-dose and 3.5 hours post-dose
  Mean temperature in degrees Celsius (°C)
Pressure Pain Threshold (PPTr) | 3.5 hours post-dose
  Mean pressure kPA
Pressure Pain tolerance threshold (PPTolTr) | 3.5 hours post-dose
  Mean pressure kPA
Peripheral nociceptor activation using Laser Doppler flowmetry | 3.5 hours post-dose
  Peripheral nociceptor activation will be assessed by monitoring cutaneous blood flow using Laser Doppler imaging
Erythema at the treated area using Erythema index | 3.5 hours post-dose
  Erythema at the treated area will be assessed using colorimetry
Stimulus-response function to graded von Frey hair stimulation | 3.5 hours post-dose
  The mean pain intensity of the stimulations on a '0-10' visual analog scale (VAS), where '0' indicates ''no pain" and '10' indicates '' the most intense pain imaginable''
Secondary pin-prick hyperalgesic area | 3.5 hours post-dose
  The area will be assessed using a 60 g weighted von Frey hair, and subjects are asked to report when the sensation changes to a "different sensation", "unpleasant" or "burning pain" sensation
Evaluation of change in body temperature | Pre-dose and up to 72 hours post-dose
  Oral temperature in degrees Celsius (˚C)

CONTACTS AND LOCATIONS:
Locations (1):
- CCBR A/S, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No